CLINICAL TRIAL: NCT04942925
Title: Clinical Comparison of Two Daily Disposable Contact Lenses - Pilot Study 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLE383-E002
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Results first posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: Myopia; Ametropia
Keywords: Contact Lenses
MeSH Terms: conditions — Myopia; Refractive Errors

STUDY DESIGN:
Intervention Model Description: Subjects will receive treatment based upon the randomized treatment sequence assignment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Precision1, then Infuse (Other): Verofilcon A contact lenses worn first, with kalifilcon A contact lenses worn second, as randomized. Each study lens type will be worn bilaterally (in both eyes) for 8 -0/+3 days in a daily disposable modality.
  Interventions: Device: Verofilcon A contact lenses; Device: Kalifilcon A contact lenses
- Infuse, then Precision1 (Other): Kalifilcon A contact lenses worn first, with verofilcon A contact lenses worn second, as randomized. Each study lens type will be worn bilaterally (in both eyes) for 8 -0/+3 days in a daily disposable modality.
  Interventions: Device: Verofilcon A contact lenses; Device: Kalifilcon A contact lenses

INTERVENTIONS:
Device: Verofilcon A contact lenses — Commercially available silicone hydrogel contact lenses for daily disposable wear
  Other Names: PRECISION1™
Device: Kalifilcon A contact lenses — Commercially available silicone hydrogel contact lenses for daily disposable wear
  Other Names: Bausch + Lomb INFUSE™

SUMMARY:
The purpose of this study is to evaluate the overall performance of PRECISION1™ contact lenses when compared to INFUSE™ contact lenses.

DETAILED DESCRIPTION:
The expected duration of subject participation in the study is up to 24 days with 3 scheduled visits.

ELIGIBILITY:
Key Inclusion Criteria:

* Able to understand and sign an Informed Consent Form that been approved by an Institutional Review Board.
* Successful wear of spherical soft contact lenses in both eyes for a minimum of 5 days per week and 10 hours per day during the past 3 months.
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Current/previous PRECISION1 or INFUSE contact lens wearer.
* Any eye condition or use of medication that contraindicates contact lens wear, as determined by the investigator.
* Routinely sleeps in contact lenses.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2021-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (4):
- United States (4):
  - Alcon Investigator 6565, Maitland, Florida
  - Alcon Investigator 6355, Orlando, Florida
  - Alcon Investigator 6583, Eden Prairie, Minnesota
  - Alcon Investigator 6313, Powell, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited from 4 investigative sites located in the United States.
Pre-assignment Details: This reporting group includes all subjects/eyes exposed to any study lenses evaluated in this study.
Units Other Than Participants: eyes
Groups:
- Precision1, Then Infuse: Verofilcon A contact lenses worn first, with kalifilcon A contact lenses worn second, as randomized. Each study lens type was worn bilaterally (in both eyes) for 8 -0/+3 days in a daily disposable modality.
- Infuse, Then Precision1: Kalifilcon A contact lenses worn first, with verofilcon A contact lenses worn second, as randomized. Each study lens type was worn bilaterally (in both eyes) for 8 -0/+3 days in a daily disposable modality.
Period: First Wear Period (8 -0/+3 Days)
Arm/Group | Precision1, Then Infuse | Infuse, Then Precision1
Started | 32; 64 eyes | 28; 56 eyes
Completed | 32; 64 eyes | 26; 52 eyes
Not Completed | 0; 0 eyes | 2; 4 eyes
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Wear Period (8 -0/+3 Days)
Arm/Group | Precision1, Then Infuse | Infuse, Then Precision1
Started | 32; 64 eyes | 26; 52 eyes
Completed | 32; 62 eyes | 26; 52 eyes
Not Completed | 0; 2 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All subjects/eyes exposed to any study lenses evaluated in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Precision1, Then Infuse | Infuse, Then Precision1 | Total
Number analyzed (Participants) | 32 | 28 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (8.2) | 35.1 (8.3) | 35.0 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 39
  Male | 11 | 10 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 28 | 28 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 27 | 23 | 50
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 32 | 28 | 60

OUTCOME MEASURES:

1. Primary Outcome: Distance VA (logMAR) With Study Lenses
Description: Distance visual acuity (VA) was assessed with study lenses in place. VA was collected for each eye separately using logarithmic of the Minimum Angle of Resolution (logMAR) charts. A logMAR acuity of 0.0 corresponds to 20/20 Snellen acuity (normal visual acuity), with a negative value denoting better than 20/20 visual acuity. No inferential testing was pre-specified for this endpoint.
Time Frame: Day 8 (-0/+3 days), each study lens type
Population: Safety Analysis Set: All subjects/eyes exposed to any study lenses evaluated in this study with non-missing response
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Groups:
- Precision1: Verofilcon A contact lenses worn bilaterally (in both eyes) during the first wear period or the second wear period, as randomized, for 8 -0/+3 days in a daily disposable modality.
- Infuse: Kalifilcon A contact lenses worn bilaterally (in both eyes) during the first wear period or the second wear period, as randomized, for 8 -0/+3 days in a daily disposable modality.
Arm/Group | Precision1 | Infuse
Number analyzed (Participants) | 58 | 58
Number analyzed (eyes) | 116 | 116
logMAR | -0.14 (0.08) | -0.15 (0.07)

ADVERSE EVENTS:
Time Frame: Adverse events (AE's) were collected from time of consent to study exit, approximately 24 days.
Description: AE's were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of participants. The safety analysis set includes all subjects/eyes exposed to any study lenses evaluated in this study.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study contact lenses
- Precision1 Ocular; Precision1 Nonocular: Events reported in this group occurred while exposed to the Precision1 contact lenses
- Infuse Ocular; Infuse Nonocular: Events reported in this group occurred while exposed to the Infuse contact lenses
Arm/Group | Pretreatment | Precision1 Ocular | Precision1 Nonocular | Infuse Ocular | Infuse Nonocular
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/116 | 0/58 | 0/120 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/116 | 0/58 | 0/120 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/116 | 0/58 | 0/120 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/25/NCT04942925/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/25/NCT04942925/SAP_001.pdf